CLINICAL TRIAL: NCT06485687
Title: Early Feasibility Study of Low-Intensity Focused Ultrasound (LIFU) Neuromodulation in Patients With Binge Eating Disorder (BED)
Brief Title: Low Intensity Focused Ultrasound for Binge Eating Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Rezai (Other)
Responsible Party: Sponsor-Investigator, Ali Rezai, Director RNI, West Virginia University
Organization: West Virginia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNI_NMD_BED01
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- LIFU Neuromodulation (Experimental)
  Interventions: Device: LIFU Neuromodulation

INTERVENTIONS:
Device: LIFU Neuromodulation — Subjects will undergo a single LIFU of the target brain region

SUMMARY:
This study is a prospective, single-center, single-arm early feasibility study, to establish safety and tolerability of LIFU for neuromodulation in patients with Binge Eating Disorder (BED)

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety, feasibility and tolerability of LIFU as an adjunct neuromodulatory treatment for BED

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females, 22 - 65 years of age.
* Participant meets DSM-5 criteria for moderate to extreme BED.
* Weight ≤450lb to accommodate in MRI.
* Shoulder width of ≤65 inches to accommodate in MRI.
* The neuromodulation targets are visible on MRI for target selection.
* Participant is able and willing to give informed consent.

Exclusion Criteria:

* Unable to undergo MR-imaging because of implanted pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent make-up or small metal fragments in the eye that welders and other metal workers may have, or if candidates are uncomfortable in small spaces (have claustrophobia).
* Participants with more than 30% of the skull area traversed by the sonication pathway are covered by scars, scalp disorders (e.g., eczema), atrophy of the scalp, or implanted objects in the skull or the brain.
* Participants with known untreated or unstable cardiac status or hypertension
* Evidence of substance (alcohol or other drug) use disorder during the previous 12 months (assessed via SCID-5).
* Past or present diagnosis of schizophrenia, psychotic disorder or bipolar disorder (assessed via SCID-5)
* Participant who is currently participating in another clinical investigation with an active treatment arm.
* Use of any medications that, in the opinion of the Investigator, may put the participant at higher risk for AEs, or impair the participant's ability to perform complete study procedures.
* Participant is considered to be a poor surgical or study candidate, which may include, but is not limited to the following: any medical, social, or psychological problem that could complicate the required procedures and evaluations of the study in the judgment of the investigator.
* Participant is pregnant/lactating or planning to be pregnant.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events | [baseline and day 7 and 90 after study procedure
  All adverse events that are related to LIFU procedure will be assessed

SECONDARY OUTCOMES:
Effect of LIFU on Food craving | Day 1, Day 7, Day 30, Day 60, Day 90; comparisons will be made relative to baseline, pre-LIFU.
  Visual Analog scale and food diary

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, Principal Investigator — WVU Rockefeller Neuroscience Institute
Locations (1):
- West Virginia University: Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States